CLINICAL TRIAL: NCT02487602
Title: A Randomized, Partially-blinded, Cross-over Scintigraphic Study to Investigate the Effect of Gelesis100 on Gastric Emptying in Overweight and Obese Subjects
Brief Title: A Scintigraphic Study to Investigate the Effect of Gelesis100 on Gastric Emptying in Overweight and Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gelesis, Inc. (Industry)
Collaborators: BDD Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: GS-100-006
Record Dates: First submitted 2015-06-26; First posted 2015-07-01 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Active Comparator): Up to 5 Gelesis100 and/or placebo capsules 30 minutes before a standard radiolabeled lunch.
  Interventions: Device: Gelesis100; Other: Placebo
- B (Active Comparator): Up to 5 Gelesis100 and/or placebo capsules 30 minutes before a standard radiolabeled lunch.
  Interventions: Device: Gelesis100; Other: Placebo
- C (Placebo Comparator): Placebo capsules 30 minutes before a standard radiolabeled lunch.
  Interventions: Other: Placebo
- D (Experimental): Up to 5 Gelesis100 and/or placebo capsules 30 minutes before a radiolabeled water.
  Interventions: Device: Gelesis100; Other: Placebo
- E (Experimental): Up to 5 Gelesis100 and/or placebo capsules 10 minutes before a radiolabeled meal.
  Interventions: Device: Gelesis100; Other: Placebo

INTERVENTIONS:
Device: Gelesis100 — Gelesis100 capsules
  Arms: A; B; D; E
Other: Placebo — Sucrose (sugar) capsules

SUMMARY:
The purpose of the study is to evaluate the gastrointestinal behaviour of a novel weight loss device in vivo to further understand the device's mechanism of action in aiding weight loss.

DETAILED DESCRIPTION:
Gelesis100 is a new, experimental medical device which has been developed by Gelesis, Inc. to aid weight loss in overweight/obese patients by reducing the amount of food required to make them feel full. The device is contained in a capsule which is swallowed with water before a meal. Once swallowed, the capsule dissolves and the capsule contents hydrate and mix with the food in the stomach, creating a feeling of fullness.

Four different treatments of up to 5 capsules each will be given to participants during this study. These will be a mixture of the Gelesis100 capsules and capsules which do not contain the device i.e., they are placebo (will contain sucrose [sugar])

The study is designed to look at:

* The time it takes for the stomach to empty once receiving each treatment
* The time it takes for food and Gelesis100 to travel through the intestine
* The effects of Gelesis100 on the feeling of satiety (how full participants feel)

In order to monitor gastrointestinal behavior, either a small amount of radioactive material will be added to a component of a standard lunch or to the water given with the treatment. The radiation emitted will then be detected as it travels through the GI tract by taking images using a device known as a gamma camera. The procedure is relatively easy and non- invasive.

ELIGIBILITY:
Inclusion Criteria:

1. Weight & Body mass index (BMI)

   1. BMI between 27 and 35 kg/m², inclusive.
   2. Body weight ≥50 kg
2. Compliance: Understands and is willing, able and likely to comply with all study procedures and restrictions.
3. Consent: Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent (signed and dated) obtained before any trial-related activities. Trial-related activities are any procedure that would not have been performed during normal management of the subject.
4. General health: Good general health with (in the opinion of the Investigator) no clinically significant and relevant abnormalities of medical history or physical examination.

Exclusion Criteria:

1. Medical History

   1. Current or recurrent disease that, in the opinion of the physician responsible, could affect the study conduct or laboratory assessments (e.g., hepatic disorders, renal insufficiency, congestive heart failure).
   2. Current or relevant previous history of serious, severe or unstable physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures.
   3. A history of current or relevant previous non self-limiting GI disorders.
   4. A history of gastric bypass or any other gastric surgery.
   5. Acute diarrhoea or constipation in the 14 days before the assessment visit. Diarrhoea will be defined as the passage of liquid faeces and/or stool frequency greater than 3 times per day. Constipation will be defined as failure to open bowels at least every other day.
   6. Currently suffering from disease known to impact gastric emptying, e.g., migraine, type 1 and type 2 diabetes.
   7. As a result of a physical examination or screening investigations, the physician responsible considers the volunteer unfit for the study.
2. Medications

   1. Subject has taken prescribed medication within 14 days prior to the first assessment visit. Subjects will be withdrawn from subsequent study days if they commence taking prescribed medication during the study period.
   2. Subject has taken over-the-counter (OTC) medication within 48 hr prior to the assessment visits. This includes the use of vitamins and natural or herbal remedies e.g., St John's Wort.
   3. Subject has taken OTC and/or prescribed Non-Steroidal Anti-Inflammatory Drugs (NSAIDS) daily or regularly within 3 months prior to the first assessment visit. Subjects will be withdrawn from subsequent study days if they commence taking OTC and/or prescribed NSAIDS during the study period.
3. Alcohol/Substance Abuse

   1. Recent history (within the last year) of alcohol or other substance abuse.
   2. Subject has an average weekly alcohol intake of greater than 21 units. 1 unit is equivalent to one 25 mL single measure of whisky, or a third of a pint of beer or half a standard (175 mL) glass of red wine.
   3. Subject has positive urine drugs of abuse test at screening.
   4. Subject has a positive breath alcohol test at screening.
4. Smoking

   1. Subject has recently discontinued smoking (less than 6 months).
   2. Subject is currently a smoker or user of nicotine-containing products.
5. Allergy/Intolerance

   1. Subject has a history of allergy to a drug, to any component of the dosage form or any other allergy, which, in the opinion of the physician responsible, contraindicates their participation.
   2. Has an allergy to any of the contents of the standardized breakfast or lunch.
   3. Subject is vegetarian.
   4. Subject is lactose intolerant.
6. Clinical Studies

   1. Participation in another clinical study (inclusive of final post-study examination) or receipt of an investigational drug within the 12 weeks before first screening visit.
   2. Previous participation in this study.
   3. Subject whose participation in this study will result in a participation in more than four studies over a 12-month period.
7. Personnel

   a. An employee of the sponsor, client or study site or members of their immediate family.
8. Radiation Exposure

   1. Subjects for whom participation in this study will exceed the limits of total radiation exposure allowed in any 12-month period (5 mSv), or will exceed 10 mSv over any three-year period.
   2. Subjects who are intending to father a child in the 3 months following the study or are unwilling to abstain from sexual intercourse with pregnant or lactating women.
   3. Subjects who are unwilling to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the assessment visit until 3 months following the study.
9. Blood

   a. Subject has donated blood or experienced significant blood loss within 3 months of screening and for the duration of the study.
10. Other a. Subject has any non-removable metal objects such as metal plates, screws etc in their chest or abdominal area.

Ages: 22 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Gastric emptying kinetics of a radiolabelled meal following administration of two different doses of Gelesis100 and placebo and two different meals | up to 10 hours on each of 3 Assessment Visit days
  Scintigraphic images of the radiation emitted by the meal will be obtained using a gamma camera. Time to 50% and 90% emptying will be assessed in addition to amount of radiation remaining in the stomach over time.
GI transit time of a radiolabelled meal following administration of two different doses of Gelesis 100 and placebo and two different meals | up to 10 hours on each of 3 Assessment Visit Days
  Scintigraphic images of the radiation emitted by the meal will be obtained using a gamma camera. Time to arrival of radiation at the colon will be assessed.

SECONDARY OUTCOMES:
Water uptake behavior of Gelesis100 | up to 10 hours on one Assesssment Visit day
  Scintigraphic images of the radiation emitted by the water will be obtained using a gamma camera. Descriptions and times related to how the radiolabelled water is taken up by Gelesis100 will be assessed.
Gastric emptying of Gelesis100 | up to 10 hours on one Assesssment Visit day
  Scintigraphic images of the radiation emitted by the water will be obtained using a gamma camera. Descriptions and times related to how the radiolabelled water empties from the stomach will be assessed.
Gastric emptying of a radiolabeled high fat meal when Gelesis100 is taken 10 minutes before the meal | up to 10 hours on one Assesssment Visit day
  Scintigraphic images of the radiation emitted by a high fat meal will be obtained using a gamma camera. Descriptions and times related to how the radiolabelled meal empties from the stomach will be assessed.
GI transit times of Gelesis100 | up to 10 hours on one Assesssment Visit day
  Scintigraphic images of the radiation emitted by the water will be obtained using a gamma camera. Time to arrival of radiation at the colon will be assessed.
GI transit times of a high fat radiolabeled meal when Gelesis100 is taken 10 minutes before the meal | up to 10 hours on one Assesssment Visit day
  Scintigraphic images of the radiation emitted by a high fat meal will be obtained using a gamma camera. Time to arrival of radiation at the colon will be assessed.
The effects of Gelesis100 on feelings of satiety | 2 hours on each of 4 Assessment Visit days
  A questionnaire will be administered several times during 2 hours on each Assessment Visit day. Area under the curve and maximum, and minimum values for the questions will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Heshmati, M.D., Study Director — Gelesis, Inc.
Locations (1):
- Bio-Images Research Ltd, Glasgow, Scotland, United Kingdom